CLINICAL TRIAL: NCT05611658
Title: Inter-observer Variation in Gross Tumor Delineation of Esophageal Cancer on MR, CT and PET CT
Status: Completed | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: 525
Record Dates: First submitted 2022-10-27; First posted 2022-11-10 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MR, PET CT — diagnostic method

SUMMARY:
The aim of the study is to investigate inter-observer variation in gross tumor volume (GTV) delineation of oesophageal cancer on different imaging modalities - CT, PET CT and MR.Twenty-three consecutive patients with esophageal cancer treated with preoperative or curative chemoradiotherapy were selected. All patients had CT, PET CT and MR imaging in treatment position prior to radiotherapy.Five experienced observers from our institution will independently delineate GTV on CT alone, MR alone, PET CT alone, on co-registered CT and MR and co-registered PET CT and MR. Inter-observer agreement, expressed in generalized conformity index (CIgen) and mean volumes of GTV will be calculated per patient and imaging modality.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced esophageal cancer eligible for treatment with preoperative or curative chemoradiotherapy

Exclusion Criteria:

* contraindications for MR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for esophageal cancer with preoperative or curative chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change of interobserver variability in target volume delineation on CT, PET CT and MR. | Through study completion, an average of 1 year.
  To compare target volume delineation of esophageal cancer using CT, PET CT and MR with determining generalized conformity indexes and mean volumes of GTV.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia